CLINICAL TRIAL: NCT05117931
Title: Phase II Study of Amivantamab in EGFR or MET- Amplified Esophagogastric Cancer
Brief Title: A Study of Amivantamab in People With Esophagogastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-324
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Esophagogastric Cancer
Keywords: metastatic; unresectable; Amivantamab; EGFR or MET amplified; 21-324
MeSH Terms: conditions — Neoplasm Metastasis | interventions — amivantamab

STUDY DESIGN:
Intervention Model Description: This is a single arm, phase II study of Amivantamab.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amivantamab (Experimental): Patients will receive amivantamab intravenously weekly for the first cycle, and biweekly subsequently at a dose of 1050mg (patients <80kg) or 1400mg (patients ≥80kg). The initial dose will be administered over 2 days in split doses in order to mitigate the risk of infusion reactions. Therapy will continue for up to 2 years or until progression of disease, initiation of alternative cancer therapy, unacceptable toxicity, or other reason to discontinue treatment occurs-whichever comes first.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Patients will receive amivantamab weekly for the first cycle, and biweekly subsequently at a dose of 1050mg (<80kg) or 1400mg (>80kg). The first day of dosing is considered Cycle 1 Day 1. Each cycle is 28 days in duration. The initial dose will be administered over 2 days to prevent infusion reactions. For patients who weigh <80 kg, amivantamab 350mg IV will be given on Cycle 1 Day 1, and the remaining 700mg IV will be given on Cycle 1 Day 2. Patients will continue to receive amivantamab 1050mg IV once a week during Cycle 1 then biweekly (Days 1 and 15) of each subsequent Cycle. For patients who weigh ≥ 80 kg, 350mg IV amivantamab will be given on Cycle 1 Day 1 and 1050mg IV will be given on Cycle 1 Day 2. Patients will continue to receive amivantamab 1400mg IV once a week during Cycle 1 then biweekly (Days 1 and 15) of each subsequent Cycle.

SUMMARY:
The purpose of this study is to see whether the study drug, amivantamab, is an effective treatment for people with EGFR- or MET-amplified esophagogastric cancer. The researchers will also look at whether amivantamab is a safe treatment that causes few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative is willing and able to provide written informed consent.
* Patients with previously treated metastatic or unresectable histologically-confirmed esophagogastric cancer who have received at least 1 line of therapy.
* EGFR or MET amplification by tissue-NGS with copy number >8 and/or ctDNA amplification by any FDA and CLIA-approved assay
* No prior receipt of an EGFR or MET inhibitor for esophagogastric cancer. (Note: if a patient previously received a EGFR inhibitor, but subsequently demonstrated a MET amplification, or previously received a MET inhibitor, but subsequently demonstrated an EGFR-amplification, inclusion is permitted).
* Patients with HER2+ (IHC 3+ or IHC 2+/FISH+) tumors must have progressed on trastuzumab.
* Measurable disease based on RECIST 1.1.
* ≥ 18 years of age on day of signing informed consent.
* Have an ECOG performance status of 0, 1, or 2.
* Adequate organ function, defined as:

A. Hemoglobin ≥9 g/dL

B. ANC ≥1.0 x 10^9 /L

C. Platelets ≥75 x 10^9 /L

D. AST and ALT ≤3 x ULN (≤5 x ULN for subjects with liver metastases)

E. Total bilirubin ≤1.5 x ULN; subjects with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits

F. Serum creatinine <1.5 x ULN or if available, calculated or measured creatinine clearance >50 mL/min/1.73 m^2

* Women of childbearing potential and male patients with women of childbearing potential partners must be willing to use an adequate method of contraception

Exclusion Criteria:

* Prior chemotherapy, targeted small molecule therapy, or biological therapy, within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (excluding alopecia).
* If subject received major surgery, they must have recovered adequately prior to starting therapy.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Known active hepatitis B (e.g., HBsAg reactive or polymerase chain reaction detectable).

Note: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.

* Known active hepatitis C (e.g., HCV RNA [qualitative] is detected).

Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.

* Other clinically active or chronic liver disease.
* Subject has uncontrolled inter-current illness, including but not limited to poorly controlled diabetes, ongoing or active infection (i.e., has discontinued all antibiotics for at least one week prior to first dose of study drug), or psychiatric illness/social situation that would limit compliance with study requirements. Subjects with medical conditions requiring chronic continuous oxygen therapy are excluded.
* Pulmonary embolism (PE) and deep vein thrombosis (DVT), within 1 month of start of study drug.
* Myocardial infarction, unstable angina, stroke, transient ischemic attach (TIA), or coronary/peripheral artery bypass graft, or any acute coronary syndrome within 6 months of start of study drug.
* Congestive heart failure defined as New York Heart Association (NYHA) Class III-IV or hospitalization for congestive heart failure (any NYHA class) within 6 months of start of study drug.
* Interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis requiring treatment with prolonged steroids or other immune suppressive agents that is unresolved or resolved within the last 3 months.
* Immune-mediated rash from checkpoint inhibitors that has not resolved prior to enrollment.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the treating investigator.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months after the last dose of trial treatment.
* Prisoners, or subjects who are compulsory detained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  ORR; defined as complete response (CR) or partial response (PR)) by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Steven Maron, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of California, Irvine, Irvine, California
  - Massachusetts General Hospital (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm